CLINICAL TRIAL: NCT05640882
Title: Is Olfaction the Key to PTSD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bar-Ilan University, Israel (Other)
Responsible Party: Principal Investigator, Sara Freedman, prof., Bar-Ilan University, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 060322sm
Record Dates: First submitted 2022-11-17; First posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-11

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VRET (Experimental): VRET - 10 week protocol using VR
  Interventions: Other: VRET
- VRET Olfaction (Active Comparator): VRET olfaction - 10 week protocol using VR with olfaction
  Interventions: Other: VRET OLFACTION

INTERVENTIONS:
Other: VRET — 10 week prolonged exposure protocol, using Virtual Reality for imaginal exposure
  Arms: VRET
Other: VRET OLFACTION — 10 week prolonged exposure protocol, using Virtual Reality for imaginal exposure with the addition of olfaction
  Arms: VRET Olfaction

SUMMARY:
Participants arriving to the ED following a potentially traumatic event such as a motor vehicle accident will be recruited into the study. Inclusion criteria: aged 18-65, Hebrew as a first language, no current psychiatric disorder. Exclusion criteria: loss of consciousness, unable to understand study procedure. Participants will answer self report questionnaires in the ED. They will be invited for a follow up interview 2 weeks and six months post trauma. Between 2 weeks and 6 months they will be folllowed up via online questionnaires. At the interviews, they will encounter 20 different olfactory stimuli, answer self-report questionnaires, and a clinical interview assessing Axis 1 disorders and PTSD will be completed. At six month, participants with PTSD will be offered therapy in the embedded RCT. Patients will receive VRET (Virtual reality exposure therapy) with or without olfaction.

DETAILED DESCRIPTION:
The goal of this project is to carry out a systematic longitudinal study with an embedded RCT examining olfactory memories in PTSD, in order to test the following hypotheses. Firstly, olfactory memories occur after all traumatic events; secondly, olfactory memories are predictors of PTSD development and thirdly, adding olfaction to PTSD treatment will enhance treatment outcome. The project comprises of a longitudinal study recruiting participants in the Emergency Room within hours of a traumatic event, assessing them at two weeks post trauma for olfactory memories, and at six months for PTSD. This will allow the first two hypotheses to be examined. Participants with PTSD and olfactory memories will be offered treatment and will be randomized to a Virtual Reality Exposure Therapy with and without added odors. Post treatment assessments will examine the third hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* hebrew native speaker
* understand study requirements

Exclusion Criteria:

* current psychiatric disorder
* suicidality
* vertigo
* epilepsy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
PTSD Status | 3 months after end of treatment
  PTSD diagnosis as measured by the CAPS
PTSD Levels | 3 months after end of treatment
  PTSD Symptoms Levels as measured by the CAPS continuous score

OTHER OUTCOMES:
PTSD Symptoms Levels Before Treatment | 6 months post traumatic event
  PTSD Symptom levels as measured by the CAPS, before treatment begins

IPD SHARING:
Plan to Share IPD: Undecided